CLINICAL TRIAL: NCT03991572
Title: Study of Individualized Accurate Targeting rTMS Intervention on Motivational Anhedonia of Treatment Resistant Depression and Brain Network Mechanism
Brief Title: rTMS Intervention on Motivational Anhedonia of Treatment Resistant Depression and Brian Network Mechanism
Acronym: rTMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Fengqiong Yu, A/Prof., Anhui Medical University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: FYu
Record Dates: First submitted 2019-04-22; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Treatment Resistant Depression; Transcranial Magnetic Stimulation; Functional Magnetic Resonance Imaging; Event-Related Potentials
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Stimulation (Active Comparator): The Real Stimulation of rTMS lasted 25 mins and delivered at 10 Hz with 1s duration,4s rest, a total of 3000 pulses at 100% of the rest motor threshold (RMT) . Behavior and MRI dataset should be acquired before the first rTMS session and after the last rTMS session.
  Interventions: Device: repeated transcranial magnetic stimulation with real coil
- Sham Stimulation (Sham Comparator): The procedure of Sham Stimulation protocol was performed by a placebo coil,lasted 25 mins and delivered at 10 Hz with 1s duration,4s rest, a total of 3000 pulses at 100% of the rest motor threshold (RMT) . MRI dataset should be acquired before the first rTMS session and after the last rTMS session.
  Interventions: Device: repeated transcranial magnetic stimulation with sham coil

INTERVENTIONS:
Device: repeated transcranial magnetic stimulation with real coil — repeated transcranial magnetic stimulation with real coil is a noninvasive technique to activate and modify the activity of the neurons
  Arms: Real Stimulation
Device: repeated transcranial magnetic stimulation with sham coil — repeated transcranial magnetic stimulation with sham coil is a placebo
  Arms: Sham Stimulation

SUMMARY:
Study of individualized accurate targeting rTMS intervention on motivational anhedonia of treatment resistant depression and brain network mechanism

DETAILED DESCRIPTION:
Before treatment, Magnetic resonance images of each participant were acquired from scanner of the same type (3.0T, Discovery GE750w). As the key role of nucleus accumbens (NACC, -7.5, 5.5, 9) in anhedonia, the accurate target of left dlPFC was defined as the strongest functional connectivity with NACC. Each treatment session was under neuronavigation with a Visor neuronavigation system (ANT Neuro, Enschede, Netherlands) for coil positioning.

All patients underwent a medical evaluation that included physical examination and routine laboratory studies before and after repetitive transcranial magnetic stimulation (rTMS) treatment. Patients were randomly allocated to real group or sham group by coin toss. A threshold of 3 points on the Hamilton Depression scale has been specified by the National Institute for Health and Care Excellence to determine a clinically meaningful difference between active pharmacotherapy and placebo. We plan to enroll minimum total sample size of 29 participants in real and sham group respectively according to the Power and Sample Size program. The decision to enroll a patient was always made prior to randomization. Patients were studied using a double-blind design. The participants, clinical raters, and all personnel responsible for the clinical care of the patient remained masked to the allocated condition and allocation parameters. Only the rTMS administrators had access to the randomization list. They had minimal contact with the patients, and no role in assessing depression. Each patient would be treated for continuous 15 days by rTMS.

Before the rTMS treatment, depression symptom of each participant was assessed by the Hamilton Depression Scale and the Beck Depression Self-Rating Scale. The anhedonia severity was evaluated by The Temporal Experience of Pleasure Scale, the Self-Report Apathy Evaluation Scale, Dimensional Anhedonia Rating Scale, the Motivation and Pleasure Scale. The neuroimaging data was collected using functional magnetic resonance imaging scan in multimodalities, resting electroencephalography, and event-related potentials during monetary incentive delay task, and Iowa-gambling test. The participants had also received a battery measure of neuropsychological tests (standardized tests to investigate their cognitive problems). After the last treatment, the same scales and neuroimaging scan were used again to assess the treatment effect of the rTMS and the underlying brain mechanism. Each participant was interviewed in detail about the adverse event of the rTMS intervention during the past 15 days. A month after the last treatment, each participant received follow-up visit by telephone to access the persistent effect of the intervention. Every participant should take part in the study in voluntary and sign an informed consent form before the study.

ELIGIBILITY:
1. Meet criteria of depression assessed by at least two psychiatrists according to the five version of Diagnostic and Statistical Manual of Mental Disorders.
2. The score of Hamilton Depression Rating Scale-24 was larger than 18.
3. The score of Montgomery-Asberg Depression Rating Scale was larger than 15.
4. Psychotropic medication was at steady dosages for at least 4 weeks prior to study entry and for the duration of the trial.
5. Age was between 18 to 60 year old.
6. The intelligence quotient score was larger than 85.
7. The education duration was at least 6 years.
8. The vision or corrected vision was normal.
9. Right handedness.
10. No treatment of rTMS, transcranial direct current stimulation or electroconvulsive therapy before.

Exclusion Criteria:

1. History of significant head trauma or neurological disorders.
2. Alcohol or drug abuse.
3. Focal brain lesions.
4. History of seizure.
5. First degree relative with epilepsy, significant neurological illness or head trauma, endocrine disease.
6. Significant unstable medical condition.
7. Recent aggression or other forms of behavioral dyscontrol.
8. Left-handedness.
9. Pregnancy.
10. Current alcohol or drug abuse
11. Inability to provide informed consent.
12. Patients with contraindications or factors affecting imaging quality, such as pacemakers, cochlear implants, or hearts Cerebrovascular metal stent, and metal denture.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Hamilton Depression Scale | baseline;15 day post-treatment
  The participants' depression symptom assessed by the Hamilton Depression Scale and the Beck Depression Self-Rating Scale change from baseline after the treatment.
Change from baseline in Motivation and Pleasure Scale | baseline;15 day post-treatment
  The severity of participants' anhedonia assessed by the Motivation and Pleasure Scale change from baseline after the treatment.

SECONDARY OUTCOMES:
The change from baseline in behavioral results of Monetary Incentive Delay task | baseline; 15 day post-treatment change from baseline after the treatment.
  The motivational anhedonia assessed by accuracy and response time in Monetary Incentive Delay task
The change from baseline in event-related brain potentials during the monetary incentive delay task | baseline; 15 day post-treatment
  The amplitudes of brain potentials of contingent negative variation, P3 and Feed-back negativity assessed by event-related brain potentials methods change from baseline after the treatment.
The change from baseline in neuroimaging results of functional magnetic resonance imaging scan in multimodalities | baseline; 15 day post-treatment
  The activation of nucleus accumbens, dorsal lateral prefrontal cortex and the functional connection these brain area assessed by functional magnetic resonance imaging scan in multimodalities change from baseline after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, MD, Study Chair — Anhui Medical University; Fengqiong Yu, MD, Study Director — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

REFERENCES:
- [Derived] Wang X, He K, Chen T, Shi B, Yang J, Geng W, Zhang L, Zhu C, Ji G, Tian Y, Bai T, Dong Y, Luo Y, Wang K, Yu F. Therapeutic efficacy of connectivity-directed transcranial magnetic stimulation on anticipatory anhedonia. Depress Anxiety. 2021 Sep;38(9):972-984. doi: 10.1002/da.23188. Epub 2021 Jun 22. PMID 34157193